CLINICAL TRIAL: NCT06057155
Title: Correlation Between Intracranial Pressure and Optic Nerve Sheath Diameter Measured With CLOSED Bundle in Patients With Acute Brain Injury: Multicenter Observational Study
Brief Title: Intracranial Pressure and Optic Nerve Sheath Diameter With CLOSED Bundle
Acronym: CLOSED
Status: Not yet recruiting | Type: Observational
Sponsor: IRCCS Istituto delle Scienze Neurologiche di Bologna (Other)
Responsible Party: Principal Investigator, Raffaele Aspide, Medical Doctor, IRCCS Istituto delle Scienze Neurologiche di Bologna
Other Study IDs: 6669
Record Dates: First submitted 2023-09-21; First posted 2023-09-28 (Actual); Last update posted 2024-03-06 (Actual); Status verified 2024-03

CONDITIONS: Intra Cerebral Hemorrhage; Subarachnoid Hemorrhage, Aneurysmal; Trauma, Brain; Hypertension Intracranial; Stroke, Ischemic
Keywords: optic nerve sheath diameter; ultrasonography; Hypertension Intracranial; neuro monitoring
MeSH Terms: conditions — Cerebral Hemorrhage; Subarachnoid Hemorrhage; Brain Injuries, Traumatic; Intracranial Hypertension; Ischemic Stroke

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (1):
- acute brain injury: Intra Cerebral Hemorrhage Subarachnoid Hemorrhage, Aneurysmal Trauma, Brain Stroke, Ischemic
  Interventions: Diagnostic Test: ultrasound optic nerve sheath diameter assessment

INTERVENTIONS:
Diagnostic Test: ultrasound optic nerve sheath diameter assessment — ultrasound optic nerve sheath diameter assessment

SUMMARY:
The design of the present study will be a multicenter prospective observational protocol. Approximately 100 patients will be recruited over the 24-month period with Acute Brain Injury (trauma brain injury, intracerebral hemorrhage, subarachnoid hemorrhage, ischemic stroke), who in their acute phase of intensive care unit require placement of a catheter capable of monitoring intracranial pressure (intra parenchymal catheter or external ventricular shunt). In addition to all the intensive care provided by the most recent guidelines, patients will undergo measurement of optic nerve sheath diameter through ultrasonography. At least, three measurements will be performed within the first 3 hours after admission, within the first 24-48 hours, and at each invasive intracranial pressure value greater than 18 cmH2O. Those patients with intracranial pressure values greater than 35 mmHg. At the first intracranial pressure measurement, patients with eyeball disease or trauma will be excluded. Measurements will be performed following the CLOSED bundle.

Analysis of the results will include correlation between the invasive pressure values and the mean value of optic nerve sheath diameter measurements in the two projections (sagittal and transverse). In addition, the correlation of the absolute value of invasive pressure detected with the ratio of the optic nerve sheath diameter measurement to the eyeball diameter measured always ultrasound will be sought.

ELIGIBILITY:
Inclusion Criteria:

acute brain injury patients with an invasive intra-cranial pressure monitoring

-

Exclusion Criteria:

patients affected by disease or trauma of eye ball patients or relatives that don't want to participate to the study

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: acute brain injury patients at risk of intra-cranial hypertension
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2024-05-01 (Estimated); Primary Completion 2025-11-01 (Estimated); Study Completion 2026-06-01 (Estimated)

PRIMARY OUTCOMES:
correlation between invasive ICP/ONSD | 3, 24, 48 hours after admission
  correlation between invasive intra-cranial pression assessment and ultasound ONSD assessment

SECONDARY OUTCOMES:
correlation between invasive intra-cranial pression assessment and ultasound ratio of ONSD assessment and eyeball transverse diameter | 3, 24, 48 hours after admission
  correlation between invasive ICP/(ONSD/ETD)

CONTACTS AND LOCATIONS:
Locations (1):
- IRCCS Istituto delle Scienze Neurologiche di Bologna, Bologna, Italy

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Background] Hansen HC, Helmke K. Validation of the optic nerve sheath response to changing cerebrospinal fluid pressure: ultrasound findings during intrathecal infusion tests. J Neurosurg. 1997 Jul;87(1):34-40. doi: 10.3171/jns.1997.87.1.0034. PMID 9202262
- [Background] Liu D, Kahn M. Measurement and relationship of subarachnoid pressure of the optic nerve to intracranial pressures in fresh cadavers. Am J Ophthalmol. 1993 Nov 15;116(5):548-56. doi: 10.1016/s0002-9394(14)73195-2. PMID 8238213
- [Background] Zoerle T, Caccioppola A, D'Angelo E, Carbonara M, Conte G, Avignone S, Zanier ER, Birg T, Ortolano F, Triulzi F, Stocchetti N. Optic Nerve Sheath Diameter is not Related to Intracranial Pressure in Subarachnoid Hemorrhage Patients. Neurocrit Care. 2020 Oct;33(2):491-498. doi: 10.1007/s12028-020-00970-y. PMID 32314244
- [Background] Vitiello L, De Bernardo M, Rosa N. Optic Nerve Sheath Diameter Evaluation With Two Ultrasound Techniques in Patients at Risk for Increased Intracranial Pressure. Crit Care Med. 2019 Sep;47(9):e787. doi: 10.1097/CCM.0000000000003811. No abstract available. PMID 31415320
- [Background] Vaiman M, Abuita R, Bekerman I. Optic nerve sheath diameters in healthy adults measured by computer tomography. Int J Ophthalmol. 2015 Dec 18;8(6):1240-4. doi: 10.3980/j.issn.2222-3959.2015.06.30. eCollection 2015. PMID 26682181
- [Background] Patterson DF, Ho ML, Leavitt JA, Smischney NJ, Hocker SE, Wijdicks EF, Hodge DO, Chen JJ. Comparison of Ocular Ultrasonography and Magnetic Resonance Imaging for Detection of Increased Intracranial Pressure. Front Neurol. 2018 Apr 24;9:278. doi: 10.3389/fneur.2018.00278. eCollection 2018. PMID 29740393
- [Background] Cochrane Central Register of Controlled Trials - Optic nerve sheath diameter as a marker of raised intracranial pressure in pediatric patients with suspected ventriculoperitoneal shunt malfunction: a pilot study Ramirez T, Abdeen N Pediatric radiology. Conference: 60th annual meeting of the society for pediatric radiology, SPR 2017. Canada, 2017, 47, S255-S256 | added to CENTRAL: 30 June 2017 | 2017 Issue 6 https://doi.org/10.1007/s00247-017-3809-x
- [Background] Robba C, Santori G, Czosnyka M, Corradi F, Bragazzi N, Padayachy L, Taccone FS, Citerio G. Optic nerve sheath diameter measured sonographically as non-invasive estimator of intracranial pressure: a systematic review and meta-analysis. Intensive Care Med. 2018 Aug;44(8):1284-1294. doi: 10.1007/s00134-018-5305-7. Epub 2018 Jul 17. PMID 30019201
- [Background] Montorfano L, Yu Q, Bordes SJ, Sivanushanthan S, Rosenthal RJ, Montorfano M. Mean value of B-mode optic nerve sheath diameter as an indicator of increased intracranial pressure: a systematic review and meta-analysis. Ultrasound J. 2021 Jul 2;13(1):35. doi: 10.1186/s13089-021-00235-5. PMID 34215966
- [Background] Aletreby W, Alharthy A, Brindley PG, Kutsogiannis DJ, Faqihi F, Alzayer W, Balhahmar A, Soliman I, Hamido H, Alqahtani SA, Karakitsos D, Blaivas M. Optic Nerve Sheath Diameter Ultrasound for Raised Intracranial Pressure: A Literature Review and Meta-analysis of its Diagnostic Accuracy. J Ultrasound Med. 2022 Mar;41(3):585-595. doi: 10.1002/jum.15732. Epub 2021 Apr 24. PMID 33893746
- [Background] Cardim D, Griesdale DE, Ainslie PN, Robba C, Calviello L, Czosnyka M, Smielewski P, Sekhon MS. A comparison of non-invasive versus invasive measures of intracranial pressure in hypoxic ischaemic brain injury after cardiac arrest. Resuscitation. 2019 Apr;137:221-228. doi: 10.1016/j.resuscitation.2019.01.002. Epub 2019 Jan 7. PMID 30629992
- [Background] Aspide R, Bertolini G, Albini Riccioli L, Mazzatenta D, Palandri G, Biasucci DG. A Proposal for a New Protocol for Sonographic Assessment of the Optic Nerve Sheath Diameter: The CLOSED Protocol. Neurocrit Care. 2020 Feb;32(1):327-332. doi: 10.1007/s12028-019-00853-x. PMID 31583527
- [Background] Aspide R, Bertolini G, Belotti LMB, Albini Riccioli L, Toni F, Mazzatenta D, Palandri G, Vetrugno L, Biasucci DG. The CLOSED protocol to assess optic nerve sheath diameter using color-Doppler: a comparison study in a cohort of idiopathic normal pressure hydrocephalus patients. Ultrasound J. 2022 Oct 29;14(1):43. doi: 10.1186/s13089-022-00291-5. PMID 36309606
- [Background] Aspide R, Bertolini G, Belotti LMB, Albini Riccioli L, Toni F, Mazzatenta D, Palandri G, Vetrugno L, Biasucci DG. Magnetic Resonance-Based Assessment of Optic Nerve Sheath Diameter: A Prospective Observational Cohort Study on Inter- and Intra-Rater Agreement. J Clin Med. 2023 Apr 5;12(7):2713. doi: 10.3390/jcm12072713. PMID 37048796
- [Background] Toms DA. The mechanical index, ultrasound practices, and the ALARA principle. J Ultrasound Med. 2006 Apr;25(4):560-1; author reply 561-2. doi: 10.7863/jum.2006.25.4.560. No abstract available. PMID 16567451